CLINICAL TRIAL: NCT02689791
Title: Effect of Resistant Wheat Starch on Subjective Appetite and Food Intake in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, James Hollis, Assistant Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: IowaSU
Record Dates: First submitted 2016-02-07; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Feeding Behavior
Keywords: Appetite; Food Intake; Satiety Hormones
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (SWF) (No Intervention): Standard Wheat Flour (SWF) Muffins
- Resistant Starch Type 4 (Experimental): Resistant Wheat Starch Muffins
  Interventions: Dietary Supplement: Resistant Starch Type 4

INTERVENTIONS:
Dietary Supplement: Resistant Starch Type 4 — single dose 26g fiber given at the breakfast meal
  Other Names: Fibersym
  Arms: Resistant Starch Type 4

SUMMARY:
A randomized, single-blind, cross-over study was conducted to determine the effect of replacing standard wheat flour (SWF) with resistant wheat starch (RWS) on markers of appetite and food intake in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-29.9 kg/m2
* Regular breakfast consumers (>5 days/week)

Exclusion Criteria:

* not weight stable (?3 kg weight change in previous 3 months)
* use/used tobacco products
* presence of acute or chronic illness
* restrained eater (>13 on the restraint section of the three-factor eating questionnaire)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Caloric intake | Single Day
  calories consumed at post-treatment lunch meal and total calories consumed on the treatment day

SECONDARY OUTCOMES:
Visual analogue scale measures of subjective appetite | Single Day
  0-100mm scale to assess hunger, fullness, thirst, desire to eat and prospective consumption
Serum concentrations of biomarkers of appetite | 150 minutes
  CCK, ghrelin, PYY3-36 and GLP-1
Plasma concentrations of biomarkers of glycemic response | 150 minutes
  Glucose, Insulin, GLP-1

IPD SHARING:
Plan to Share IPD: Undecided